CLINICAL TRIAL: NCT03945617
Title: Optimizing Psychotherapy for Anxiety Disorders
Acronym: OPTIMAX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: Psychiatric University Hospital, Zurich (Other); Swiss National Science Foundation (Other); University of St.Gallen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10001C_169827
Record Dates: First submitted 2018-07-27; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Anxiety Disorders
Keywords: anxiety; cognitive behavior therapy; transdiagnostic treatment; prediction
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This is randomized controlled trial involving a before-after design with an intervention group that receives immediate access to treatment and a waitlist-control group.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded regarding treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unified treatment protocol (Experimental): This intervention group receives 16 sessions of CBT-based, individual psychotherapy using to the Unified Treatment Protocol for the treatment of emotional disorders by Barlow et al. (2011).
  Interventions: Behavioral: Unified Treatment Protocol
- Waitlist Control Group (No Intervention): Participants in the waitlist control group gain access to the Unified Treatment after a waiting period of 16 weeks

INTERVENTIONS:
Behavioral: Unified Treatment Protocol — The Unified Treatment Protocol (UP) is a transdiagnostic psychotherapeutic treatment manual for emotional disorders, that is based on CBT principles and focuses on changing dysfunctional emotion regulation.
  Arms: Unified treatment protocol

SUMMARY:
Anxiety disorders are highly prevalent and are associated with a high burden of disease, costs and individual impairment worldwide. Psychotherapy, especially cognitive behavioral therapy (CBT), is the first line treatment for anxiety disorders. CBT is effective in modifying dysfunctional cognitions and reducing avoidance behavior, thus leading to a lasting reduction of symptoms.

Even though CBT is generally effective, around 50% of patients do not benefit sufficiently from this treatment. The current study aims at optimizing the treatment of anxiety disorders by identifying predictors of treatment response. Multiple (neuro-)psychological, biological, genetic and behavioral variables will be combined into a comprehensive prediction model of treatment outcome. Knowledge on predictors can then be used to improve therapy on an individual patient level.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18-65 years
* one of the following primary axis I disorders according to the Diagnostic and Statistical Manual of Mental Disorders (DSM): Panic Disorder with or without Agoraphobia; Social Anxiety Disorder; Anxiety Disorder not otherwise specified, Adjustment Disorder with Anxiety, Adjustment Disorder with Mixed Anxiety and Depression; Specific Phobia; Generalized Anxiety Disorder
* if on medication If on medication or in other types of treatments, patients must be willing to remain stable on their treatment for the duration of the acute phase/therapy of the study
* not currently receiving other psychotherapeutic treatment for anxiety or another condition
* fluent German
* provision of written informed consent

Exclusion Criteria:

* concomitant psychotherapy
* medical relative contraindications involve conditions that impede thorough exposure, e.g. cardiovascular diseases, autoimmune diseases or pregnancy
* current or past schizophrenia, psychosis, or bipolar disorder
* current suicidal ideation.
* current substance/alcohol dependence or abuse
* cluster A or B personality disorder
* pregnancy (for women)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale | change from T0 (entry to study) at mid-treatment (8 weeks after T0), change from T0 at post-treatment (after 16 weeks from T0), change from T0 at 6 months follow-up and change from T0 at one year from post-treatment
  clinician rating of anxiety symptoms, range: 0-56, with higher values representing a worse outcome
Overall Anxiety Severity and Impairment Scale | change from T0 (entry to study), at mid-treatment (8 weeks after T0), change from T0 at post-treatment (16 weeks after T0), change from T0 at 6 months follow-up and change from T0 at one year post-treatment
  self-report measure of anxiety symptom severity and impairment; range: 0-20, with higher values representing worse outcome

SECONDARY OUTCOMES:
Hamilton Depression Scale | change from T0 (entry to study), at mid-treatment (8 weeks after T0), change from T0 at post-treatment (16 weeks after T0), change from T0 at 6 months follow-up and change from T0 at one year post-treatment
  clinician rating of depressive symptoms; range: 0-66, with higher values representing worse outcome
Beck Depression Inventory | change from T0 (entry to study), at mid-treatment (8 weeks after T0), change from T0 at post-treatment (16 weeks after T0), change from T0 at 6 months follow-up and change from T0 at one year post-treatment
  self report measure of depression; range: 0-63, with higher values indicating worse outcome
Social Functioning Index (SFI) | change from T0 (entry to study), at mid-treatment (8 weeks after T0), change from T0 at post-treatment (16 weeks after T0), change from T0 at 6 months follow-up and change from T0 at one year post-treatment
  change in social functioning; Subscales: "work" (range: 1-15) and "leisure time" (range: 1-30), with higher numbers indicating worse outcome
World Health Organization-5 Wellbeing Index | change from T0 (entry to study), at mid-treatment (8 weeks after T0), change from T0 at post-treatment (16 weeks after T0), change from T0 at 6 months follow-up and change from T0 at one year post-treatment
  change in well-being; range: 0-25, with higher values indicating a better outcome
Beck Anxiety Inventory | change from T0 (entry to study), at mid-treatment (8 weeks after T0), change from T0 at post-treatment (16 weeks after T0), change from T0 at 6 months follow-up and change from T0 at one year post-treatment
  self-report in anxiety symptoms, range 0-63, with higher values representing worse outcome

OTHER OUTCOMES:
Test of self-conscious affect | change from T0 (entry to study), at mid-treatment (8 weeks after T0), change from T0 at post-treatment (16 weeks after T0), change from T0 at 6 months follow-up and change from T0 at one year post-treatment
  self-report to index self-conscious affect; 3 subscales: shame self-talk, guilt self-talk, blaming others; each ranging from 0 to 55, with higher values indicating a worse outcome
Thought Control questionnaire | change from T0 (entry to study) at mid-treatment (8 weeks after T0), change from T0 at post-treatment (16 weeks after T0), change from T0 at 6 months follow-up and change from T0 at one year post-treatment
  self-report measure to assess worry and reappraisal as cognitive strategies/information processing; subscales "worry" (range: 1-24, with higher values indicating worse outcome) and "reappraisal" (range:1-24, with higher values representing better outcome) are reported

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Kleim, Prof. Dr., Principal Investigator — University of Zurich
Locations (1):
- University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Muller-Bardorff M, Schulz A, Paersch C, Recher D, Schlup B, Seifritz E, Kolassa IT, Kowatsch T, Fisher A, Galatzer-Levy I, Kleim B. Optimizing Outcomes in Psychotherapy for Anxiety Disorders Using Smartphone-Based and Passive Sensing Features: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 May 14;13:e42547. doi: 10.2196/42547. PMID 38743473